CLINICAL TRIAL: NCT01389986
Title: Effects of Gum Chewing on Recovery of Bowel Function Following Abdominal Surgery for Endometrial and Ovarian Cancer: a Randomized Controlled Trial
Brief Title: Effects of Gum Chewing on Recovery of Bowel Function Following Abdominal Surgery for Endometrial and Ovarian Cancer
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kittipat Charoenkwan, MD, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GUM-ET/OV
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Paralytic Ileus
MeSH Terms: conditions — Intestinal Pseudo-Obstruction | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gum chewing (Experimental): Gum chewing (30 minutes in duration each time, 4 times/days at the usual time of meal, until the first flatus) in addition to conventional postoperative feeding schedule
  Interventions: Behavioral: Gum chewing
- Conventional (No Intervention): Conventional postoperative feeding schedule

INTERVENTIONS:
Behavioral: Gum chewing — Gum chewing (30 minutes in duration each time, 4 times/days at the usual time of meal, until the first flatus) in addition to conventional postoperative feeding schedule
  Arms: Gum chewing

SUMMARY:
Following extensive abdominal surgery for the treatment of endometrial or ovarian cancer, paralytic ileus frequently develops. Gum chewing can promotes the return of bowel function through the cephalic-vagal reflex and increased intestinal enzymes secretion.

The objectives of this study are to evaluate effects of adding gum chewing to the conventional postoperative feeding protocol on the return of bowel function, its related complications, and patients' satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing staging or cytoreductive surgery for primary endometrial or ovarian cancer at Maharaj Nakorn Chiang Mai hospital

Exclusion Criteria:

* Perioperative hyperalimentation
* Recent chemotherapy (within 3 weeks before surgery)
* Previous bowel surgery
* Inflammatory bowel diseases
* Previous abdominal or pelvic radiation
* Need for immediate postoperative endotracheal intubation
* Need for postoperative admission to intensive care unit
* Undergoing emergency surgery with oral intake of fluid or food within 4 hours before surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Time to first flatus | Up to 7 days after surgery

SECONDARY OUTCOMES:
Incidence and severity of postoperative nausea, vomiting,and abdominal discomfort | Up to 7 days after surgery
Incidence of postoperative complications | Up to 7 days after surgery
Time to first regular diet | Up to 7 days after surgery
Time to first defecation | Up to 7 days after surgery
Postoperative analgesics requirement | Up to 7 days after surgery
Hospital stay | On the day of hospital discharge, an expected average of 7 days
Patients' satisfaction | Up to 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Kittipat Charoenkwan, MD, Principal Investigator — Chiang Mai University
Locations (1):
- Faculty of Medicine, Chiang Mai University, Chiang Mai, Chiang Mai, Thailand